CLINICAL TRIAL: NCT00337922
Title: Post-Marketing Clinical Study of EPZICOM Tablet (Lamivudine / Abacavir Sulfate) - Pharmacokinetic Study in HIV-Infected Patients -
Brief Title: Pharmacokinetic Study Of EPZICOM Tablet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104807
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infection
Keywords: EPZICOM; Lamivudine; Abacavir; pharmacokinetics; Japanese
MeSH Terms: conditions — HIV Infections | interventions — abacavir, lamivudine drug combination

INTERVENTIONS:
Drug: Lamivudine / Abacavir Sulfate

SUMMARY:
This study was designed to explore the drug levels in the blood in Japanese HIV-infected patients taking EPZICOM tablet at least for 2 weeks prior to administration of the study drug. Pharmacokinetics after administration of EPZICOM tablet will be investigated in a total of 8 subjects.

ELIGIBILITY:
Inclusion criteria:

* A Japanese HIV-infected patient who continues to use one EPZICOM tablet in the morning (00:00 to 12:00) at least for 2 weeks prior to administration of the study drug.
* A patient who agrees to abstain from alcohol from 48 hours prior to administration of the study drug until completion of blood sampling for pharmacokinetic analysis.

Exclusion criteria:

* A patient developing AIDS (Patients who developed AIDS in the past but have no symptoms or findings that may serve as indicators at screening may be eligible for the study.)
* A patient with a history of hypersensitivity to the study drug and the ingredients (lamivudine, abacavir sulfate) of the study drug

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8
Dates: Start 2006-07

PRIMARY OUTCOMES:
The following pharmacokinetic parameters of plasma lamivudine and abacavir Maximum plasma concentration(Cmax), Time to the maximum plasma concentration(tmax), Elimination half-life(t1/2), Area under the plasma concentration-time curve(AUC)

SECONDARY OUTCOMES:
Safety (adverse events occurring during the study period)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (4):
- Japan (4):
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo